CLINICAL TRIAL: NCT01663909
Title: The Efficacy of Guided Imagery on Pain, Anxiety, and Coping for Adolescents Post-spinal Fusion
Brief Title: Pain Management Using Guided Imagery for Adolescents Post-spinal Fusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Sylvie Charette, Clinical Nurse Specialist, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Scoliosis
Record Dates: First submitted 2012-06-27; First posted 2012-08-13 (Estimated); Last update posted 2012-08-13 (Estimated); Status verified 2012-08

CONDITIONS: Pain; Scoliosis
Keywords: Pain; Scoliosis; Rehabilitation; Cognitive-behavioral interventions; Adolescents
MeSH Terms: conditions — Pain; Scoliosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (No Intervention)
- Guided imagery (Experimental)
  Interventions: Behavioral: Guided imagery intervention

INTERVENTIONS:
Behavioral: Guided imagery intervention — A 30-min DVD was developed which included general information on pain management as well as a section on guided imagery using sounds and images.
  Arms: Guided imagery

SUMMARY:
Surgery to correct scoliosis (spinal fusion)generates a severe pain intensity rending pain management a complex task. Several studies have found out that pharmacological interventions alone were not enough to provide optimal pain management for these patients. The investigators developed a DVD on guided imagery, customized for teenagers, to help them cope better with their pain. The investigators believe that this type of intervention combined with their usual analgesic medication will help them to control their pain and foster rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 11 and 20 years old
* Have undergone a posterior/anterior arthrodesis surgery for idiopathic scoliosis
* Able to write and understand French
* Requires a computer or DVD player at home.

Exclusion Criteria:

* Diagnosed with a moderate cognitive deficit or severe mental retardation

Ages: 11 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Actual)
Dates: Start 2010-05; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Level of pain intensity | Level of pain intensity at two weeks after the surgery
  Pain was measured before the patients left the hospital on their 7th postoperative day (T-1, time of discharge from hospital). It was measured again at two week post-discharge (T-2) and also at one month post-discharge (T-3) on their visit to the orthopedic clinic. Our primary outcome was at T-2.

SECONDARY OUTCOMES:
Level of anxiety | Level of anxiety from 24-hrs before the surgery, to two weeks and to one month after the surgery
  Anxiety was measured as baseline data on the pre-operative visit (24 hrs before surgery). It was also measured at two weeks post-discharge and at one month on the day of the visit to the orthopedic clinic.
Level of coping | Level of coping from Baseline (pre-operative), to two weeks and to one month after the surgery
  Coping strategies of adolescents regarding their pain management were also measured pre-operatively (24 hrs before surgery), at two weeks and one month post-surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvie Le May, RN, PhD, Study Director — Université de Montréal
Locations (1):
- CHU Ste-Justine Hospital, Montreal, Quebec, Canada